CLINICAL TRIAL: NCT05862441
Title: A Study to Assess the Efficacy of Omnivirol-Salicylic Acid Combination Therapy for Cutaneous Warts With Emphasis on Persistent Warts
Acronym: OVW-SA001
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Nina Redzic, Study Coordinator, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OVW-SA001
Record Dates: First submitted 2023-04-23; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Cutaneous Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AV2-SA (Experimental): 100% AV2 (v/v) - 17% SA (w/v) treatment one drop daily and 10% AV2 (v/v) spray one puff weekly
  Interventions: Drug: AV2-SA2
- SA (Active Comparator): 100% d-carvone (v/v) - 17% SA (w/v) treatment one drop daily and 10% d-carvone (v/v) spray one puff weekly
  Interventions: Drug: SA

INTERVENTIONS:
Drug: AV2-SA2 — AV2 is a combination of FDA GRAS-label approved organic compounds (natural essential oils: carvone, eugenol, geraniol, and nerolidol) that is postulated to be able to prevent viral entry and proliferation by deactivating the infectious virions before they enter the cell. Salicylic acid (SA) formulations are the most commonly used preparations in the treatment of warts. SA is an organic acid that destroys epidermal cells and softens hyperkeratotic epidermis. Implementation of AV2-SA combination therapy would ensure permanent lesion clearance by on the one hand inactivation of HPV by AV2, and on the other hand elimination of the lesion by SA treatment.
  Arms: AV2-SA
Drug: SA — Salicylic acid (SA) formulations are the most commonly used preparations in the treatment of warts. SA is an organic acid that destroys epidermal cells and softens hyperkeratotic epidermis.
  Arms: SA

SUMMARY:
Cutaneous warts comprise an extremely common condition caused by infection with the human papillomavirus (HPV). Although most verrucae will disappear spontaneously, many patients do seek treatment. Current wart treatments do not target the cause of the lesion directly, resulting in variable treatment efficacies and high wart recurrence rates. AV2 is a broad-spectrum antiviral drug, that is capable of deactivating HPV. It is however not able to destruct the already infected cells, which raises the need for an additional ablative treatment i.e. salicylic acid (SA). Implementation of AV2-Salicylic acid (AV2-SA) combination therapy would ensure permanent lesion clearance by on the one hand inactivation of HPV by AV2, and on the other hand elimination of the lesion by SA treatment. The primary aim of this study is to assess the efficacy of AV2-SA treatment versus standard SA treatment, by comparing cure and recurrence rates of cutaneous warts between the two treatment groups (at 12 weeks and six months after randomization). The second aim is to assess the safety and tolerability of AV2-SA therapy. The third aim is to identify subgroups of cutaneous warts that have favorable response to treatment, by comparing cure rates in an HPV genotype-specific manner. This randomized controlled trial will enroll 260 participants with cutaneous warts who will either receive the AV2-SA combination therapy or SA control treatment. Real time monitoring will be possible by daily photographs sent via WhatsApp TM (a messaging application) as well as online follow-up questionnaires administered on several occasions. HPV genotyping will be performed on swab self-samples.

ELIGIBILITY:
Inclusion Criteria:

* Must exhibit one or more cutaneous warts.
* Must agree to refrain from using prescription or supplemental antiviral medications without first obtaining permission of the attending healthcare professional.
* Must be 12 years or older.
* Must be able to read Dutch.
* Must be willing to sign informed consent.
* Must be willing and able to self-assess and use WhatsApp, a freely available messaging application, for follow-up.

Exclusion Criteria:

* Exhibits only seborrheic and/or facial warts. Salicylic acid treatment is not suitable for facial warts. Seborrheic warts are not caused by HPV infection.
* Is immunocompromised.
* Has already participated in another clinical trial concerning treatment for cutaneous warts within six months before enrollment in this study or currently is in a trial evaluating other treatments for his/hers warts.
* Has a medical history of any severe diseases like hepatitis, renal or liver dysfunction, cardiovascular, gastrointestinal, malignant tumors, or psychiatric disorders, etc., which might influence the assessments or conduct of the trial by the discretion of the investigator.
* Has known or suspected allergic or adverse response to the investigational product AV2, its components or salicylic acid.
* Has impaired healing or neuropathy, for example owing to diabetes, peripheral vascular disease or any other condition.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of AV2-SA treatment versus standard SA treatment: cure rate | 12 weeks after enrollment
  To assess the efficacy of AV2-SA treatment versus standard SA treatment by comparing cure rates of the index warts between the two treatment groups at 12 weeks after enrollment.
Efficacy of AV2-SA treatment versus standard SA treatment: recurrence rate | 6 months after enrollment
  To assess the efficacy of AV2-SA treatment versus standard SA treatment by comparing recurrence rates of the index warts between the two treatment groups at 6 months after enrollment.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events in the AV2-SA treatment group versus the standard SA treatment group. | 12 weeks after enrollment
  The safety of both treatments will be assessed by monthly questionnaires actively asking the participants if they experienced any pain or other treatment-related adverse events. Pain will be measured with a scale of 1 to 4, with score 1 representing no pain at all and score 4 extreme pain.
To compare time to clearance of index wart between the two treatment groups | 6 months after enrollment
To compare change in size of index wart between the two treatment groups | 6 months after enrollment
To compare number of verrucae remaining between the two treatment arms | 6 months after enrollment
To determine the genotype-specific distribution of wart-associated HPV types in a Belgian population (according to the age, wart location, postal code, etc.) | through study completion, an average of 1 year
To investigate the prevalence of mucosal HPV types in cutaneous warts | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Redzic N, Pereira AR, Menon S, Bogers J, Coppens A, Kehoe K, Vanden Broeck D. Characterization of type-specific HPV prevalence in a population of persistent cutaneous warts in Flanders, Belgium. Sci Rep. 2023 Oct 15;13(1):17492. doi: 10.1038/s41598-023-44154-y. PMID 37840107